CLINICAL TRIAL: NCT01825824
Title: Multicenter Phase II Study of Stereotactic Ablative Radiotherapy for Hepatocellular Carcinoma ≤ 5 cm
Brief Title: Stereotactic Ablative Radiotherapy for Hepatocellular Carcinoma ≤ 5 cm
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korea Cancer Center Hospital (Other)
Collaborators: Dongnam Institute of Radiological & Medical Sciences (Other); Soonchunhyang University Hospital (Other); Inje University (Other); Inha University Hospital (Other); Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Mi-Sook Kim, Doctor, Korea Cancer Center Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-1205-001-005; KCT0000454 (Registry Identifier: Clinical Research information Service); KROG 12-02 (Registry Identifier: Korean Radiation Ocology Group); K-1205-001-005 (Other: Korea Institute of Radiological & Medical Science IRB)
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Stereotactic ablative radiotherapy; Stereotactic body radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic ablative radiotherapy (Experimental): Stereotactic ablative radiotherapy for unresectable hepatocellular carcinoma with size ≤ 5 cm and 3cm apart from gastrointestinal tract after incomplete trans-arterial chemo-embolization
  Interventions: Radiation: Stereotactic ablative radiotherapy

INTERVENTIONS:
Radiation: Stereotactic ablative radiotherapy — The HCC patients with size ≤5 cm and 3 cm apart from gastrointestinal tract will be included in this study. Total stereotactic ablative radiotherapy (SABR) doses will be 60 Gy in 3 fractionations. Patients receive 3 fractionations separated by >48 hours. At least 700 ml of normal liver (entire liver minus cumulative GTV) should not receive a total dose of > 17 Gy in three fractions. If volume of normal liver does not exceed 700 ml, at least 70% of normal liver should not receive a total dose of > 17 Gy. Dose of esophagus, stomach and intestine do not exceed 30 Gy.
  Other Names: Stereotactic body radiotherapy

SUMMARY:
The standard treatment for hepatocellular carcinoma (HCC) is surgery, such as, by hepatic resection or liver transplantation, but less than 20% of HCC patients are suitable for surgery. In the remaining patients with inoperable and advanced HCC, trans-arterial chemo-embolization (TACE) has been widely used but TACE alone rarely produces complete response and commonly develops recurrence. Recently several small studies reported high tumor response and local control rate after stereotactic ablative radiotherapy (SABR) alone or with TACE for inoperable HCC. This study will evaluate SABR effect with 60 Gy in 3 fractionations for HCC with size of ≤ 5 cm and 3 cm apart from gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 20 years of age
* Initially diagnosed or recurrent hepatocellular carcinoma (HCC)
* Unresectable HCC
* Cirrhotic status of Child Pugh class A or B7
* Eastern Cooperative Oncology Group performance status 0 or 1
* single or sum of multiple tumor ≤ 5 cm
* HCC with 3 cm apart from gastrointestinal tract
* The volume of uninvolved must be at least 700 ml
* Incomplete response after trans-arterial chemo-embolization of 1-5
* A single lesion or multiple lesions including portal vein tumor thrombosis included in radiation field with one or consecutive sessions of stereotactic body radiation therapy (SBRT)
* No evidence of an uncontrolled lesion at any other site
* No evidence of complications of liver cirrhosis
* No evidence of uncontrolled inter-current illness
* Patient or guardian must be able to provide verbal and written informed consent

Exclusion Criteria:

* Patient with previous history of abdominal radiation
* Direct invasion to esophagus, stomach or colon by HCC

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Local control rate | up to 1 year
  From the date of SABR to the date of local failure or last follow-up

SECONDARY OUTCOMES:
Overall survival rate | up to 2 years
  From the date of SABR to the date of death or last follow-up
Progression free survival rate | up to 2 years
  From the date of SABR to the date of first failure or last follow-up
Intrahepatic recurrence free survival rate | up to 2 years
  From the date of SABR to the date of Intrahepatic recurrence or last follow-up
Treatment related toxicity | up to 1 year
  Adverse events using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0; Classic radiation induced liver disease; Non-classic Classic radiation induced liver disease; Worsening of Child-Turcotte-Pugh score; Worsening of MELD score

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Sook Kim, MD, PhD, Principal Investigator — Korea Cancer Center Hospital, Korea Institute of Radiological and Medical Sciences
Locations (7):
- South Korea (7):
  - Inje University Haeundae Paik Hospital, Busan
  - Dongnam Institute of Radiological & Medical Sciences, Busan
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Catholic University Incheon St. Mary's Hospital, Incheon
  - Inha University Hospital, Incheon
  - Korea Cancer Center Hospital, Korea Institute of Radiological and Medical Sciences, Seoul
  - Soon Chun Hyang University Hospital Seoul, Seoul

IPD SHARING:
Plan to Share IPD: Undecided